CLINICAL TRIAL: NCT02328989
Title: Pessary to Prevent Prematurity in Twins in Case of Short Cervix
Acronym: PESSAR'ONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13 7048 01
Record Dates: First submitted 2014-10-01; First posted 2014-12-31 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2020-07

CONDITIONS: Pregnancy
Keywords: prematurity; short cervix; twin pregnancy; pessary
MeSH Terms: conditions — Premature Birth | interventions — Pessaries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pessary (Experimental): The device will be placed in the vagina during the consultation. It is rinsed in sterile water for lubrification and left in place until delivery or remove at 36 weeks in case of no delivery before. There is no need to use any analgesia. The good position of the pessary is checking in the same time than the placement with digital examination.
  Interventions: Device: Pessary
- No pessary (No Intervention): No pessary will be placed in the vagina.

INTERVENTIONS:
Device: Pessary — The device will be placed in the vagina during the consultation. It is rinsed in sterile water for lubrification and left in place until delivery or remove at 36 weeks in case of no delivery before. There is no need to use any analgesia. The good position of the pessary is checking in the same time than the placement with digital examination.
  Arms: Pessary

SUMMARY:
For 25 years, the twin pregnancy rate has regularly increased in the majority of European countries and in the United States, by 35% between 1981 and 2006. Increased use of medically assisted procreation and older maternal age are the two main causes. At the present time twin pregnancies represent nearly 20% of premature deliveries. The rate of very premature births (< 32-34 weeks) is 7 times higher in twin pregnancies than in singleton pregnancies. As prematurity accounts for 75% of neonatal morbidity and mortality, and extreme prematurity is the principal cause of neonatal mortality and of brain sequelae in twins, the search for a preventive treatment appears as a priority in perinatal medicine. The investigators recently showed in a prospective multicenter study that cervical ultrasound at 22 and 27 wks was a better predictive investigation of premature delivery < 34 wks than digital examination. Recently in a randomized trial in a population of short-cervix singleton pregnancies, the premature delivery rate decreased by 40% in the pessary group compared with the usual management group. No other trial of pessary use in short-cervix twin pregnancies was published today. Recently, in a historical comparison of twins with twin-to-twin transfusion syndrome treated with laser, Carreras et al. have showed a decreased rate of preterm delivery with the use of pessary in case of short cervix. The investigators wish to set up a randomized multicenter study in France in the population of short-cervix twin pregnancies to show a potential benefit of the pessary compared with simple surveillance.

DETAILED DESCRIPTION:
For 25 years, the twin pregnancy rate has regularly increased in the majority of European countries and in the United States, by 35% between 1981 and 2006. Increased use of medically assisted procreation and older maternal age are the two main causes. At the present time twin pregnancies represent nearly 20% of premature deliveries. The rate of very premature births (< 32-34 weeks) is 7 times higher in twin pregnancies than in singleton pregnancies. As prematurity accounts for 75% of neonatal morbidity and mortality, and extreme prematurity is the principal cause of neonatal mortality and of brain sequelae in twins, the search for a preventive treatment appears as a priority in perinatal medicine. The investigators recently showed in a prospective multicenter study that cervical ultrasound at 22 and 27 wks was a better predictive investigation of premature delivery < 34 wks than digital examination.[1] As there is currently no recommended preventive treatment for prematurity in twin pregnancies[2], the 2009 guidelines of the College of Obstetricians leave the teams with the option of carrying out systematic cervical ultrasound or not during follow-up investigations.[3] Recently in a randomized trial in a population of short-cervix singleton pregnancies, the premature delivery rate decreased by 40% in the pessary group compared with the usual management group.[4] In a recent multicenter trial (ProTWIN), while therapeutic efficacy of the pessary (versus usual management) was not demonstrated in the overall group of twin pregnancies, in the short-cervix subgroup (< 25th percentile of the population) the < 32 wks delivery rate decreased from 29% to 14% (OR= 0.49 (0.24-0.97) and neonatal morbidity also decreased.[5] No other trial of pessary use in short-cervix twin pregnancies was published today. Recently, in a historical comparison of twins with twin-to-twin transfusion syndrome treated with laser, Carreras et al. have showed a decreased rate of preterm delivery with the use of pessary in case of short cervix.[6] The investigators wish to set up a randomized multicenter study in France in the population of short-cervix twin pregnancies to show a potential benefit of the pessary compared with simple surveillance.

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic twin pregnancies between 16 and 24+0 weeks CL < 25th percentile for GA

- < 35mm between 16 and 24+0d weeks Vaginal swabs for bacteriological analysis < 72 hours Patient age > 18 years Written informed consent obtained French first language (speak, read, understand) French social security cover

Exclusion Criteria:

* Painful regular contractions
* Major fetal abnormalities
* Fetal malformation
* Active vaginal bleeding, placenta praevia
* Discordance fetal weight more than 40%
* Treatment with progesterone
* Patient with cerclage
* Ruptured of membrane
* Twin to twin transfusion syndrome
* Uterine malformation
* Chronic maternal disease (diabetes, hypertension, renal insufficiency, Heparin Treatment)
* Conisation history
* patients subject to a judicial safeguard order, participating in another research study including an exclusion period which has not expired at the time of screening will not be included

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2014-11; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
perinatal death or significant neonatal morbidity until discharge from the hospital | 6 months
  it's a composite outcome : perinatal death (i.e medical interruption of pregnancy, intrauterine fetal death, or death occurring during the first four weeks after birth, before day 29), or significant neonatal morbidity until discharge from the hospital, defined as one or more of the following complications: bronchopulmonary dysplasia (BPD), intraventricular haemorrhage (IVH) grade III or IV, periventricular leucomalacia (PVL), necrotizing enterocolitis (NEC) grade II or higher, culture proven sepsis, retinopathy of prematurity (ROP) requiring treatment.

SECONDARY OUTCOMES:
Preterm delivery | 6 months
To evaluate the prolongation of pregnancy in days | 6 months
The differential cost-efficacy ratio of the two strategies | 6 months
Tolerance of the pessary | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Vayssière, PhD, Study Director — University Hospital, Toulouse
Locations (18):
- France (18):
  - CHU Toulouse, Toulouse, France
  - CHRU Lille, Lille, Lille
  - Hôpital Saint-Joseph, Marseille, Marseille
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - Hôpital Marseille AP-HM, Marseille
  - CHU Nantes, Nantes
  - GH Pitié Salpétriêre, Paris
  - Hôpital Antoine Béclère, Paris
  - Hôpital Bicêtre, Paris
  - Hôpital Necker, Paris
  - Hôpital Robert Debré, Paris
  - Maternité Port-Royal Cochin, Paris
  - CHI Poissy, Poissy
  - CHU Saint-Etienne, Saint-Etienne
  - Hôpital Universitaire de Strasbourg, Strasbourg
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Groussolles M, Winer N, Sentilhes L, Biquart F, Massoud M, Vivanti AJ, Bouchghoul H, Rozenberg P, Olivier P, Desbriere R, Chauleur C, Perrotin F, Coatleven F, Fuchs F, Bretelle F, Tsatsaris V, Salomon LJ, Sananes N, Kayem G, Houflin-Debarge V, Schmitz T, Benoist G, Arnaud C, Ehlinger V, Vayssiere C; Groupe de Recherche en Gynecologie Obstetrique. Arabin pessary to prevent adverse perinatal outcomes in twin pregnancies with a short cervix: a multicenter randomized controlled trial (PESSARONE). Am J Obstet Gynecol. 2022 Aug;227(2):271.e1-271.e13. doi: 10.1016/j.ajog.2022.01.038. Epub 2022 Feb 3. PMID 35123930